CLINICAL TRIAL: NCT02287818
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL OF AC-201 IN SUBJECTS WITH GOUT
Brief Title: A Study of AC-201 Controlled-Release Tablet (CR Tablet) in Patients With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-201-GOU-002
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — diacerein; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo plus Febuxostat
  Interventions: Drug: Placebo; Drug: Febuxostat
- AC-201 (Experimental): AC-201 CR tablet plus Febuxostat
  Interventions: Drug: AC-201; Drug: Febuxostat

INTERVENTIONS:
Drug: Placebo — Placebo twice daily from Day 1 to Week 12
  Other Names: PBO
  Arms: Placebo
Drug: AC-201 — AC-201 CR tablet 100 mg twice daily from Day 1 to Week 12
  Other Names: AC-201 CR tablet
  Arms: AC-201
Drug: Febuxostat — Febuxostat 40 mg once daily from Week 4 to Week 16; titration to 80 mg once daily at Week 8 as needed to achieve serum uric acid concentration <6 mg/dL
  Other Names: ULT

SUMMARY:
The study is designed to test the urate-lowering effect, safety, and tolerability of AC-201CR in an initial dosing period, followed by the addition of a ULT to test the efficacy and safety of the combination and prophylaxis of gout flares during ULT.

DETAILED DESCRIPTION:
AC-201CR is a control released formulation of AC-201 that in previous clinical studies showed potential dual effects in both reducing serum uric acid (sUA) and gout flares. The mechanism of action of AC-201 includes the inhibition of the production and activity of caspase-1 and interleukin-1β (IL-1β), and selective inhibition of re-absorption transporters in the kidney. The goal of gout treatment is to reduce serum uric acid (sUA) concentrations below the urate solubility limit while avoiding acute gout flares. However, the initiation of urate-lowering therapy (ULT) increases the occurrence of acute gouty arthritis flares. IL-1β plays a key role in mediating this inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 20 to 65 years, inclusive.
2. Meets ≥6 of the 12 American College of Rheumatology preliminary criteria (1977) for the classification of acute arthritis of primary gout (Appendix 2), OR have proven tophus or documented monosodium urate (MSU) crystals in the joint fluid.
3. Serum uric acid ≥7.5 mg/dL and ≤10 mg/dL at screening with ≥1 gouty arthritis flare within one year prior to screening, OR serum uric acid ≥9 mg/dL and ≤10 mg/dL at screening with or without prior gout flares.

Exclusion Criteria:

1. Use of allopurinol, febuxostat, benzbromarone, probenecid, or sulfinpyrazone within 2 weeks prior to screening.
2. Occurrence of a gouty arthritis flare within 1 week prior to screening or during the screening period through baseline.
3. Use of colchicine within 1 week prior to screening.
4. Use of Glucocorticoids, NSAIDs or COX-2 inhibitors within 1 week prior to screening.
5. Allergy, contraindication, or intolerance to febuxostat.
6. Severe renal impairment.
7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) concentration >2 times the upper limit of laboratory normal range (>2x ULN) at screening.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Youh Tsai, Principal Investigator — Taipei Veteran General Hospital (TVGH)
Locations (1):
- Taipei Veteran General Hospital (TVGH), Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | AC-201
Started | 60 | 67
Completed | 53 | 54
Not Completed | 7 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AC-201 | Total
Number analyzed (Participants) | 60 | 67 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.1) | 47.3 (11.7) | 47.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 59 | 62 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 60 | 67 | 127
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 60 | 67 | 127

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Serum Uric Acid Concentration <6.0 mg/dL
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AC-201
Number analyzed (Participants) | 60 | 67
Participants | 33 | 43

ADVERSE EVENTS:
Arm/Group | Placebo | AC-201
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/67
Other Adverse Events (participants affected / at risk) | 29/60 | 43/67
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | AC-201 (N=67)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 0
Cardiac disorders (Cardiac disorders) | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 7 | 25
General disorders and administration site (General disorders) | 1 | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 2
Immune system disorders (Immune system disorders) | 0 | 1
Infections and infestations (Infections and infestations) | 5 | 6
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 0
Investigations (Investigations) | 6 | 6
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 6 | 6
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nervous system disorders (Nervous system disorders) | 1 | 4
Renal and urinary disorders (Renal and urinary disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin And subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 1
Vascular disorders (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes